CLINICAL TRIAL: NCT02022293
Title: Atorvastatin in Preventing Nasopharyngeal Carcinoma Patients Receiving Radiotherapy From Carotid Stenosis: A Multicenter, Double-blind, Placebo-Controlled, Randomized Trial
Brief Title: Atorvastatin in Preventing Nasopharyngeal Carcinoma Patients Receiving Radiotherapy From Carotid Stenosis
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment target could not be achieved.
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professer, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2013018; SYSN003
Record Dates: First submitted 2013-12-11; First posted 2013-12-27 (Estimated); Last update posted 2017-12-04 (Actual); Status verified 2017-12

CONDITIONS: Nasopharyngeal Carcinoma; Radiation Therapy Complication
Keywords: Nasopharyngeal Carcinoma; Radiotherapy; Carotid Stenosis; Atorvastatin
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Carotid Stenosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Atorvastatin (Active Comparator): Patients will take atorvastatin 20mg per night, totally 2 years.
  Interventions: Drug: Atorvastatin
- Placebo (Placebo Comparator): Patients will take placebo once per night for 2 years. The appearance and dosage of placebo will be the same as atorvastatin.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Atorvastatin — Patients in this group will take 20mg per night.
  Other Names: Atorvastatin Calcium Tablets; Lipitor
  Arms: Atorvastatin
Other: Placebo
  Arms: Placebo

SUMMARY:
Patients with head and neck cancer who underwent irradiation have a higher risk of developing severe carotid stenosis, and eventually develop to transient ischemic attack or stroke. However, it's still not clear whether early intervene in vascular risk factors is benefit for patients after radiotherapy.

Our study aimed to evaluate the feasibility and safety of atorvastatin for preventing NPC patients after radiotherapy from severe carotid stenosis. In a randomized, double-blind, placebo-controlled trial, about 324 nasopharyngeal carcinoma (NPC) patients will be enrolled from six centers in Guangdong Province and randomized 1:1 to atorvastatin group or placebo group.

DETAILED DESCRIPTION:
It is a randomized, double-blind, placebo-controlled trial, about 324 nasopharyngeal carcinoma (NPC) patients will be enrolled from six centers in Guangdong Province and randomized 1:1 to atorvastatin group (20mg per night, totally 2 years) or placebo group. All Patients will be followed up for 2 years. Ultrasound and Transcranial Color Doppler (TCD) will be used to evaluate the changes of intima-media thickness (IMT) and occurrence of plaque formation of carotid arteries. Safety will be monitored every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have received radiation therapy for histologically confirmed nasopharyngeal carcinoma.
* Prior irradiation <3 years prior to study entry.
* Male or fertile women who are willing to take contraception during the trial.
* Age 40-65 years old.
* Carotid stenosis < 50%.
* LDL-C between 100mg/dL（2.5mmol/L）and 190mg/dL（4.9mmol/L）.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of bleeding related to tumor or radiotherapy during or after radiation.
* Evidence of tumor invasion to major vessels(for example the carotid artery).
* Severe complications, such as history of stroke, myocardial infarction, liver diseases, thyroid dysfunction, inadequately controlled hypertension and epilepsy.
* Familial hypercholesterolemia.
* Taking lipid-lowing drugs.
* Aspartate aminotransferase(AST) or alanine aminotransferase(ALT) >upper limits of normal (ULN), creatinine >ULN.
* Allergic history of atorvastatin.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in maximal of IMT of bilateral carotid arteries | At baseline and 2 years
  Patients will take Ultrasound and Transcranial Color Doppler every 6 months to measure the thickness of intima-media thickness (IMT) and occurrence of plaque formation of carotid arteries. We will compare the maximal IMT of bilateral carotid arteries at 2 years from baseline.

SECONDARY OUTCOMES:
Incidence of sever carotid stenosis | At 2 years
  Patients will be followed up for 2 years. We defined sever carotid stenosis as stenosis>50% by using ultrasound and TCD.
Incidence of cardiovascular events | At 2 years
  Patients will be followed up for 2 years and cardiovascular events such as stroke, transient ischemic attack (TIA) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Peng, Ph.D, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (6):
- China (6):
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zengcheng People's Hospital, Licheng, Guangdong
  - The Affiliated Hospital of Guangdong Medical College, Zhanjiang, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi